CLINICAL TRIAL: NCT03029195
Title: Efficacy of Nasoalveolar Molding Therapy for Treatment of Unilateral Cleft Lip and Palate in Egyptian Infants
Brief Title: Nasoalveolar Molding for Egyptian Cleft Lip Palate Infants
Acronym: EgyCleft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mona Sabry Mostafa Saad, Lecturer of Prosthodontics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlexandriaU
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Cleft Lip Palate; Cleft Lip, Unilateral, Complete
Keywords: cleft lip and palate; nasoalveolar molding; Egyptian infants; quantitative analysis
MeSH Terms: conditions — Cleft Lip | interventions — Nasoalveolar Molding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study group (Experimental): Nasoalveolar molding therapy for cleft lip and palate infants
  Interventions: Device: Nasoalveolar molding therapy
- Control group (No Intervention): No nasoalveolar molding therapy for cleft lip and palate infants
- Age matched Norms (No Intervention): Normal (non-cleft) age matched infants

INTERVENTIONS:
Device: Nasoalveolar molding therapy — Presurgical infant orthopedics
  Arms: Study group

SUMMARY:
The cleft lip and palate (CLP) is the commonest craniofacial anomaly worldwide. Nasoalveolar molding (NAM) therapy has emerged in the management of CLP as an early presurgical intervention to provide symmetry to severely deformed nasal cartilage, achieve projection to the flattened nasal tip, provide nonsurgical elevation for the columella, improve alignment of the alveolar ridge, reduce the cleft gap and it could significantly reduce the number of secondary surgeries. Despite that NAM therapy is becoming the treatment option for early cleft care, there is growing debate about its efficacy due to lack of quantitative assessment of these findings. To provide the highest levels of clinical evidence on NAM therapy, there has been international call for Randomized Controlled Clinical Trials.

Statement of the problem: lack of quantitative data about the efficacy of the NAM therapy for unilateral CLP.

Aim of the study: is to develop a standardized non-invasive quantitative assessment for two different techniques of the NAM therapy in Egyptian infants that involves 3D laser scanning/CAD analysis for maxillary geometry, and nasal anthropometric analysis.

Methods Trial design: Prospective randomized controlled clinical trial (RCT). Settings: The RCT will be performed through two phases; (Phase I: A controlled pre and post-RCT that will be designed for the quantitative evaluation of the NAM therapy on the maxillary geometry), and (Phase II: A post-test RCT will be designed for the quantitative evaluation of the NAM therapy on the nasal anthropometry and comparing the outcome with the nasal anthropometry that will be performed to age matched Egyptian norms).

Participants: 30 Egyptian infants with nonsyndromic UCLP will be randomly allocated to study groups (Group I, n=15) that will undergo NAM therapy before the primary surgical repair, and control group (n=15) that will undergo the primary surgical repair without NAM therapy. And 15 Egyptian infants will act as norm group.

Follow-up: (phase I- T0: before NAM, T1: after 1 month and T2: before surgery). (Phase II- T"0: 10 days after surgery, and T"1: 6 months after surgery).

DETAILED DESCRIPTION:
o Trial Design:

The present randomized controlled clinical trial (RCT) will be performed through two phases:

• RCT- (Phase I)

A controlled pre- and post-clinical trial will be designed for the quantitative evaluation of the NAM therapy on the maxillary geometry.

• RCT- (Phase II)

A post-test controlled clinical trial will be designed for the quantitative evaluation of the NAM therapy on the nasal anthropometry.

Infants with nonsyndromic complete unilateral cleft lip and palate UCLP will be selected from those admitted to the Maxillofacial and Plastic surgery department- Faculty of Dentistry- Alexandria University based on the inclusion and exclusion criteria.

* Sample size:

Using a power of 80% to detect clinically meaningful difference at the cleft gap distance (D1-D2) before and after applying NAM therapy = 5.8, SD (standard deviation) =3.4, effect size=1.2 and α=0.05. The minimal required sample size was calculated to be twelve per group (increased to fifteen to avoid drop outs).

The sample size was calculated using G*Power software.

o Randomization:

The randomization for a total of 45 infants will be done as following:

Thirty infants with nonsyndromic UCLP will be randomly allocated by using closed envelop allocation concealment method. However, the fifteen normal infants will be only randomly selected.

RCT- (Phase I)

o Study group

(Group I): 15 infants In this group infants will undergo presurgical nasoalveolar molding before the primary surgical correction

o Control group

(Group II): 15 infants This group, the infants will undergo primary surgical correction without presurgical NAM procedures.

RCT- (Phase II)

* Norm group: (Group III): 15 infants Age matched noncleft infants. A group of normal age matched noncleft infants will be randomly selected to act norms for the nasal anthropometry for the Egyptian model, and will be compared with will be compared with the study and the control groups.

  • Procedures and Measurements:
  1. Procedures

     RCT- (Phase I)

     1.1. Case history, examination, and diagnosis

     1.2. Impressions and working cast:

     Following evaluation and a thorough explanation of the treatment goals and the procedure to the parents, an impression of an intraoral cleft defect will be made using fast setting alginate impression material loaded on a custom made tray made from wax.

     With the infant fully awake and without any anesthesia in a clinical setting prepared to handle an airway emergency with a surgeon present as a part of the impression team.

     During impression making, the infant will be held in an inverted position to keep the tongue forward and to allow fluids to drain out of the oral cavity.

     Once the impression material has been set, the tray will be removed, and the oral cavity will be examined for the residual impression material in the cleft region.

     Intraoral impressions will be carefully poured in regular dental stone, and the casts will be recovered carefully.

     1.3. Fabrication of the appliance:

     The fabrication of the NAM appliance will be done following the technique described by Grayson et al. It includes an intraoral molding acrylic palatal plate and a nasal stent.

     All casts will be marked and stored for measurements.

     • The oral molding appliance:

     The cleft region of the palate and alveolus will be filled in with wax to approximate the contour and topography of an intact arch. The cast will be duplicated to obtain a working cast on which two layers of wax will be adapted and laboratory processed using clear heat-cure acrylic resin to fabricate the molding prosthesis of 2 to 3 mm thickness to provide structural integrity and to permit adjustments during the molding therapy.

     The appliance will be finished and polished to ensure that all tissue borders are smooth and that the oral portion of the appliance that would be in contact with the dorsum of the tongue is given a high polish.

     At the insertion appointment, the appliance will be carefully fitted in the infant's oral cavity and observed for few minutes. The infant should able to suckle without gagging or struggling.
     * Extraoral retentive button:

     An extraoral retentive button will be fabricated with self polymerizing clear acrylic resin (*) and positioned facing downward on the labial flange, at an angle 40◦ relative to the plate, allowing clearance for upper and lower lips that will facilitate the positive seating of the appliance to the palatal tissues.

     The appliance will be then secured extraorally to the cheeks and bilaterally by surgical tapes with orthodontic elastics at each end.

     The use of skin barrier dressing tapes will be advocated to reduce cheek irritation.
     * Retentive taping with adhesive tapes and orthodontic elastics:

     The skin barrier dressing tapes will be first applied to the infant's cheeks, lateral and superior to the commissure.

     These base tapes will also serve to anchor the thinner (0.25 × 4 inch) tapes of suture strips used to hold the appliance against the palate.

     Small orthodontic elastics (inner diameter 0.25 inch, wall thickness heavy) will be incorporated into the loops of thinner tapes folded over them.

     The elastic band will be placed over the retentive button, and the thinner tapes will be pulled and secured to the base tapes on the infant's cheeks posteriorly and superiorly.

     An additional broader tape will be applied over the ends of the thinner tapes to anchor suture strips and elastic bands to the base tapes.

     The parents will be provided with detailed instructions on the proper method of lip taping along with taping materials and adhesive. The patient will be recalled on a weekly basis for follow-up.

     Before any adjustments, the appliance will be cleaned with soap and water. Adhesive tapes and elastics will be changed every week to maintain the proper activation force to mold the alveolar segments. Instructions will be given to keep the appliance in the oral cavity for 24 hours except during cleaning. The tissue surface of the appliance will be modified to allow selective pressure on the greater and lesser alveolar segments on either side of the cleft for correct alignment.
     * Nasal stent

     Within the first month of treatment, the phase of active nasal cartilage molding begins when the intraalveolar gap reduced to approximately 6 mm by incorporation of the nasal stent component.

     A nasal stent will be constructed from 0.019 inch round stainless steel wire. It will be extended forward and then curved backward in the form of a "swan neck" entering 3 to 4 mm past the nostril aperture.

     Finally, the superior aspect of the nasal stent will be covered with a thin layer of soft liner to ensure positive elastic pressure to the internal tissues of the nasal dome.

     The upper lobe will be inserted into the nose and gently lifted toward the dome until a moderate amount of tissue blanching is evident. The lower lobe of the nasal stent will lift the nostril apex and define the top of the columella. Periodic examination of the tissues and adjustment of the appliance will be continued every week to mold the nasoalveolar complex into the desired shape and position.

     The endpoint for the treatment of patients with NAM will be when the inter-segment distance will have been less than 3 mm and the nasal cartilages, columella, and philtrum will have been properly repositioned, ensuring a clinically desirable approximation of the alveolar segments.

     The infant will scheduled for surgical repair with the plastic surgeon after parents' consent.

     1.4. Weekly adjustment visits

     Weekly adjustments are required for maximum effectiveness of the presurgical appliance. On each visit, a new impression will be taken and poured with dental stone. This will be done to examine cleft closure and guide adjustment to the appliance modifications. . Sporadic emergency appointments are also needed to resolve any ulceration which may develop.

     RCT- (Phase II)

     1.5. Surgery

     The primary surgical closure of the lip and nose will be performed at 3 months of age.

     The surgical technique will be performed according to Millard's rotation/advancement technique. Because the alveolar segments will be in approximation, a gingivoperiosteoplasty will be performed.

     Digital photos with a submento-vertical view will be taken to the infants face after the surgical closure. ( T"0 = 10 days post-surgery) and (T"1= 6 months post-surgery).
  2. Measurements:

     2.1. Quantitative 3D maxillary geometric analysis.

     2.2. Quantitative nasal anthropometric analysis on photographs. (Photogrammetry).

     RCT- (Phase I)

     2.1. Quantitative 3D maxillary geometric analysis:

     The impressions for the maxillary casts that would have been taken at the initial visit (T0; pre-NAM therapy), (T2 during NAM therapy) and (T3 before surgery) will undergo 3D laser scanning and computer aided design (CAD) analysis.

     The 3D models will be constructed using a laser scanning machine (3Shape) and 3D software for CAD analysis.

     Reference points and lines, which are based on the anatomic structures, will be identified and digitized on the 3D model. The linear, angular, midline deviation, distance, and curvature of the arch will be identified.

     After laser scanning, the reference base plane will be set by. The plane containing the points located at the incisal point (A) and the tuberosity points on the noncleft and cleft sides (T1, T2) defined the XY-plane (horizontal reference plane).

     On the 3D image, the outline of the upper alveolar arch will be marked using six points that contained the anatomical landmarks (D1, A, C1, M1, and T1 on the major segment and D2, C2, M2, and T2 on the minor segment).

     The curvature radius of the appropriate circle of the upper alveolar arch on each major and minor segment (R and r, respectively) will be calculated using the software.

     The symmetry of the upper alveolar arch will be analyzed by calculating the ratio of the curvatures of the upper alveolar arch on the major and minor segments (R/r ratio) by using the following formula: R/r ratio = the curvatures of the appropriate circle of the upper alveolar arch on the major segment (R)/the curvatures of the appropriate circle of the upper alveolar arch on the minor segment (r). The R/r ratios at the time of lip and palatal repair will be compared between the NAM and non-NAM groups.

     RCT- (Phase II)

     2.2. Quantitative nasal anthropometric analysis on photographs (Photogrammetry):

     Comparing the affected and unaffected sides after surgery by direct digitization process of the nasal morphology after surgical repair through quantifying the geometry of the nasal cavity.

     Digital photographs will be taken after the primary surgical repair for the infants head to obtain submento-vertical views including the recommended landmarks. Landmarks, constructs and reference lines anthropometric landmarks on face and nose will be selected as extracted from the geometrical condition of the discriminated nostril coordinates.

     The algorithm aims to simplify the process of extracting Area Of Interest (AOI), in our case is the face, extracting Region(s) Of Interest (ROI), in our case are the eyes, nose, etc.

     There are two main steps:

     I- Pre-processing steps:
     1. This is about identifying the AOI through Image threshold where face boundaries are identified.
     2. Within AOI, facial features are identified such as eyes to be used as reference points to define the horizontal baseline.
     3. Vertical symmetry axis is identified as the perpendicular line on horizontal baseline passing through the mid point between eyes.

        II- Processing steps:
     4. Get nose data (ROI).
     5. Mirror the normal side.
     6. Mark the difference between the normal and actual state.
     7. Calculate statistics and geometrical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian infants.
* Infants should present with nonsyndromic complete UCLP ,
* Infant age should be less than 90 days.
* The infant's family agreed to undergo NAM therapy.

Exclusion Criteria:

* Congenital malformations and soft tissue bands.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Three dimensional (3D) change in the maxillary geometry. | (T0 baseline; pre-NAM therapy), (T2 during NAM therapy) and (T3 before surgery)
  CAD analysis for the maxillary casts that will be obtained from the cleft infants in both study and control group.

SECONDARY OUTCOMES:
Change in the nasal anthropometry. | ( T"0 = 1 days post-surgery) and (T"1= 6 months post-surgery).
  Photogrammetric analysis for photographs that will be taken for the cleft infants in both study and control group.

OTHER OUTCOMES:
Nasal anthropometry of age-matched (6 months old) Egyptian norms. | ( T"0 = 10 days post-surgery) and (T"1= 6 months post-surgery).
  Photogrammetric analysis for photographs that will be taken for the age-matched norm group.
  anthropometry with the Egyptian norms

CONTACTS AND LOCATIONS:
Overall Officials: Mona S. Saad, MSc, Principal Investigator — Alexandria University
Locations (1):
- Faculty of dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grayson BH, Santiago PE, Brecht LE, Cutting CB. Presurgical nasoalveolar molding in infants with cleft lip and palate. Cleft Palate Craniofac J. 1999 Nov;36(6):486-98. doi: 10.1597/1545-1569_1999_036_0486_pnmiiw_2.3.co_2. PMID 10574667
- [Background] Braumann B, Keilig L, Bourauel C, Jager A. Three-dimensional analysis of morphological changes in the maxilla of patients with cleft lip and palate. Cleft Palate Craniofac J. 2002 Jan;39(1):1-11. doi: 10.1597/1545-1569_2002_039_0001_tdaomc_2.0.co_2. PMID 11772163
- [Background] Clark JM, Skoner JM, Wang TD. Repair of the unilateral cleft lip/nose deformity. Facial Plast Surg. 2003 Feb;19(1):29-40. doi: 10.1055/s-2003-39134. PMID 12739180
- [Background] Meara JG, Andrews BT, Ridgway EB, Raisolsadat MA, Hiradfar M. Unilateral cleft lip and nasal repair: techniques and principles. Iran J Pediatr. 2011 Jun;21(2):129-38. PMID 23056779
- [Background] Sommerlad BC. International confederation for cleft lip and palate and related craniofacial anomalies task force report: palatoplasty in the speaking individual with unrepaired cleft palate. Cleft Palate Craniofac J. 2014 Nov;51(6):e122-8. doi: 10.1597/14-124. Epub 2014 Jul 9. PMID 25007031
- [Background] Singh GD, Levy-Bercowski D, Santiago PE. Three-dimensional nasal changes following nasoalveolar molding in patients with unilateral cleft lip and palate: geometric morphometrics. Cleft Palate Craniofac J. 2005 Jul;42(4):403-9. doi: 10.1597/04-063.1. PMID 16001922
- [Derived] Saad MS, Fata M, Farouk A, Habib AMA, Gad M, Tayel MB, Marei MK. Early Progressive Maxillary Changes with Nasoalveolar Molding: Randomized Controlled Clinical Trial. JDR Clin Trans Res. 2020 Oct;5(4):319-331. doi: 10.1177/2380084419887336. Epub 2019 Dec 20. PMID 31860800